CLINICAL TRIAL: NCT06889740
Title: A Prospective, Multi-center, Double-blind, Placebo-controlled, Randomized, Multiple-arm, Parallel Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of UthPeak NMNH (Reduced Nicotinamide Mononucleotide) in Healthy Adult Participants
Brief Title: Evaluate the Safety, Tolerability, and Efficacy of UthPeak NMNH (Reduced Nicotinamide Mononucleotide) in Healthy Adult Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EffePharm LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Study No. EP_RNM_001_24
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Healthy Aging
Keywords: UthPeak; NMNH; reduced NMN; reduced nicotinamide mononucleotide

STUDY DESIGN:
Intervention Model Description: Multi-center, Double-blind, Placebo-controlled, Randomized, Multiple-arm, Parallel Study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Placebo Comparator): Ingredient: Starch Dosage form: Capsule, 125mg/capsule Frequency: 2 capsules per day Duration: 90 days
  Interventions: Other: Placebo
- Group 2 (Experimental): Ingredient: NMNH Dosage form: Capsule, 62.5 mg/capsule Frequency: 2 capsules per day Duration: 90 days
  Interventions: Other: NMNH
- Group 3 (Experimental): Ingredient: NMNH Dosage form: Capsule, 125 mg/capsule Frequency: 2 capsules per day Duration: 90 days
  Interventions: Other: NMNH
- Group 4 (Experimental): Ingredient: NMNH Dosage form: Capsule, 250 mg/capsule Frequency: 2 capsules per day Duration: 90 days
  Interventions: Other: NMNH

INTERVENTIONS:
Other: NMNH — Reduced Nicotinamide Mononucleotide
  Arms: Group 2; Group 3; Group 4
Other: Placebo — Starch powder
  Arms: Group 1

SUMMARY:
This study is to assess the safety and tolerability of NMNH as a dietary supplement for human consumption. The current study aims to comprehensively evaluate its potential effects on pharmacokinetics, physical performance, biological age and overall quality of life. These findings will expand our understanding of NMNH therapeutic potential and guide its future clinical applications in anti-aging interventions.

DETAILED DESCRIPTION:
A total of 80 healthy adult participants were considered for enrolment in the study based on predefined eligibility criteria and screening assessments, which included demographics, medical history, clinical laboratory tests, diagnostic evaluations, and prior medication review.

The 80 participants were randomly assigned to placebo group, NMNH 125 mg group, NMNH 250 mg group, or NMNH 500 mg group, and oral supplementation for 90 consecutive days.

Baseline assessments comprised NAD+ levels, BMI, biological age evaluation, a six-minute walking test, and a quality-of-life assessment. These parameters were also evaluated during Day 45 and day 90 . Participants were formally enrolled in the study after reconfirmation of eligibility.

Blood samples were collected at multiple time points (0h, 0.5h, 1h, 2h, 4h, 6h, 12h, and 24h) after the first dose of supplementation to assess NAD+ levels. Pharmacokinetic parameter assessments were conducted exclusively for the second set of 10 participants in each group who provided informed consent.

Throughout the study, physical examinations, vital signs, concomitant medications, and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy male/females aged 40 to 65 years.
2. Participants with Body Mass Index (BMI) between 18.5 and 35 kg/m2.
3. Participants who are willing to provide written Informed Consent for participating in the study
4. Participants who are able to follow verbal and written study directions.
5. Participants must be able to maintain consistent diet and lifestyle habits throughout the study.
6. Participants must be willing to agree to use effective contraceptive methods while on treatment and for 3 months after the completion of study.
7. Participants willing to administer assigned dietary supplements for 3 months.

Exclusion Criteria:

1. Participants on current use of prescription or over-the-counter nicotinic acid.
2. Participants using any statin drugs.
3. Participants having used any tobacco product or used a recreational drug in the past 6 months.
4. Participants having abnormal screening laboratory test values or other lab test result(s) that would preclude study participation in the judgment of the investigator.
5. Participants with documented presence of atherosclerotic disease and/or cardiopulmonary disease.
6. Participants with history of drug or alcohol abuse.
7. Participants with history of unstable depression or mental illness within the last 6 months for which the investigator believes could impact the participant's ability to comply with study requirements.
8. Participants unwilling to discontinue use of conventional multivitamin/mineral or other supplements at least two weeks prior to the start of study.
9. Participants who are currently participating in or planning to begin a weight loss diet during the study period.
10. Participants who chronically use over-the-counter medication which would interfere with study endpoints.
11. Participants whose lifestyle or schedule incompatible with the study protocol.
12. Participants with known hypersensitivity to the drug components used during the study.
13. Female participants with positive result for urinary beta human chorionic gonadotropin or gestation period or breastfeeding.
14. Other diseases or medications, according to the investigator, that would interfere directly in the results of the study or jeopardize the health of the participant.
15. Currently, or within the past 30 days, enrolled in a different clinical investigation.
16. Inability to provide a venous blood sample.
17. Unable or unwilling to provide written informed consent for participation in study.
18. Patients with a current diagnosis of any form of cancer within the past 5 years, regardless of disease stage or treatment status, are ineligible for participation in this clinical trial. Any history of cancer within this timeframe must be documented and confirmed through medical records or pathology reports.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
To assess NAD+ Values in blood | day 0, day 45, day 90
  To assess NAD+ Values in blood
Assessment of Biological Age | day 0, day 45, day 90
  Assessment of Biological Age by an online biological age calculator
Physical Performance walking test | day 0, day 45, day 90
  Physical Performance is assessed by endurance test measured on six minutes
Change in BMI | day 0, day 45, day 90
  BMI
Quality (QoL) Questionnaire | day 0, day 45, day 90
  The 36-Item Short Form Health Survey (SF-36) was used to assess Health-Related Quality of Life. It measures eight scales: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores range from 0 to 100, with higher scores indicating a more favorable health state.

SECONDARY OUTCOMES:
Safety will be assessed based on number of adverse events | day 0, day 45, day 90
  Safety will be assessed based on number of adverse events
Tolerability will be assessed based on number of subjects drop out due to treatment related adverse events | day 0, day 45, day 90
  Tolerability will be assessed based on number of subjects drop out due to treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Li, Study Director — EffePharm LTD
Locations (2):
- India (2):
  - Medstar Speciality Hospital, Bengaluru, Karnataka
  - Vinayaka Mission's Medical College and Hospital, Kāraikāl, Puducherry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zapata-Perez R, Tammaro A, Schomakers BV, Scantlebery AML, Denis S, Elfrink HL, Giroud-Gerbetant J, Canto C, Lopez-Leonardo C, McIntyre RL, van Weeghel M, Sanchez-Ferrer A, Houtkooper RH. Reduced nicotinamide mononucleotide is a new and potent NAD+ precursor in mammalian cells and mice. FASEB J. 2021 Apr;35(4):e21456. doi: 10.1096/fj.202001826R. PMID 33724555
- [Background] Smolin AG. Ab Initio Studies of NMNH(2-) Conformers in Water-Methanol Solutions: Comparative Analysis of the Biexponential Fluorescence Signals for NMNH(2-) and NADH. J Phys Chem B. 2022 Dec 29;126(51):10870-10881. doi: 10.1021/acs.jpcb.2c08220. Epub 2022 Dec 16. PMID 36524597